CLINICAL TRIAL: NCT03482908
Title: Evaluating Coordination of Care Between Pediatricians and Women Infants & Children (WIC) Nutritionists: Early Obesity Prevention for WIC Mothers and Children
Brief Title: Coordination of Care Between Pediatricians and Women Infants & Children Nutritionists
Acronym: WEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency); Geisinger Clinic (Other); Pennsylvania Bureau of Women, Infants & Children (WIC) (Unknown)
Responsible Party: Principal Investigator, Jennifer Savage Williams, Assistant Professor of Nutritional Sciences, Penn State University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1 R40MC283170100
Record Dates: First submitted 2018-03-23; First posted 2018-03-29 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Childhood Obesity
Keywords: Responsive parenting
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: A multi-site, randomized controlled trial (RCT) to test that hypothesis that an individually tailored responsive parenting obesity prevention intervention that coordinates care provided by WIC nutritionists and primary care providers will be effective to ultimately reduce/prevent obesity in infants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Responsive parenting treatment (Experimental): Early Healthy Lifestyles (EHL) screening tool reported by participants to identify potentially obesogenic parenting practices and child behaviors; data sharing/coordination into electronic health records to inform counseling by trained providers; responsive parenting curriculum delivered by trained WIC nutritionists.
  Interventions: Behavioral: Early healthy lifestyles; Behavioral: Responsive parenting curriculum; Behavioral: Data sharing/coordination
- Standard Care Control (No Intervention): Standard of pediatric and WIC care

INTERVENTIONS:
Behavioral: Early healthy lifestyles — Patient reported data to identify parenting practices and child behaviors associated with child's obesigenic risk in the future
  Other Names: EHL
  Arms: Responsive parenting treatment
Behavioral: Responsive parenting curriculum — Information from the American Academy of Pediatrics Healthy Active Living for Families (HALF) program supplemented with messages from the INSIGHT study, that were written at the 5th grade reading level, with messages focused on 4 categories: 1) feeding the baby 2) soothing the baby 3) sleep health and 4) playing with the baby
  Arms: Responsive parenting treatment
Behavioral: Data sharing/coordination — Data integration into child's electronic health record that is shared between settings (WIC and GHS PCPs) with display and documentation features that informs counseling.
  Arms: Responsive parenting treatment

SUMMARY:
WEE Baby Care is a 6 month intervention that coordinates care across multiple settings- health care clinics and WIC clinics on responsive parenting practices to increase parenting competence thereby preventing infant rapid weight gain. The investigators will recruit mother/infant dyads in Central PA, who participate in the Women, Infants, and Children (WIC) program and receive clinical care from a Geisinger pediatrician participating in this study.

DETAILED DESCRIPTION:
This multi-site, randomized, controlled trial (RCT) will test the hypothesis that an individually tailored responsive parenting obesity prevention intervention that coordinates care provided by WIC nutritionists and primary care providers (PCPs) will be more effective than usual care at 1) delivering consistent messages and 2) changing maternal and infant behavior to 3) reduce/prevent rapid infant growth from birth to 6 months.

Geisinger research staff will recruit mother/infants dyads primarily from newborn nurseries from Geisinger Health Systems hospitals in Central Pennsylvania (PA). Mother-infant dydas may also be recruited directly from newborn well-child visits, prenatal WIC visits, and using social media platforms such as Facebook. Key eligibility criteria include that infants participate in the Special Supplemental Women, Infants and Children (WIC) program and receive clinical care from a participating Geisinger Health Systems pediatrician. Upon eligibility and receiving consent, mother/infant dyads will be randomized to 1 of 2 groups: intervention (coordination of care) or control (Geisinger standard of pediatric care), stratified on infant birth weight, race, and parity. In this study, coordination of care is defined at two levels: (1) PCPs and WIC will deliver the same, consistent messages and (2) providers will communicate with each other on preventive care plans regarding responsive parenting and nutrition education.

The intervention will consist of 3 components: 1) a parent self-assessment and screening survey called Early Healthy Living/Lifestyles (EHL) tool to assess the child's future obesity risk and tailor education; 2) parenting and nutrition education using the Healthy Active Living for Families curriculum (HALF) developed by the American Academy of Pediatrics, supplemented by evidence-based materials that teach mothers alternatives to using feeding to manage infant behavior, and establishing good sleep hygiene; and 3) coordination of care between PCPs and WIC nutritionists utilizing HIT. Components 1 and 2 focus on teaching mothers to recognize hunger and fullness signs in their infants, use alternative soothing strategies to feeding, develop good sleep hygiene routines, and engage in active social play.

Once consented and enrolled, all parents receive a welcome packet with brief parenting tips tailored to the group assignment. Intervention participants will also be mailed the responsive parenting curriculum after enrolling that addresses the domains of infant sleep, feeding, soothing and play. Pediatricians who have patients enrolled and randomized to the intervention group will have access to the EHL data in the patient's electronic health record which they then use to record notes about each well child visit. After each well-child visit, these notes including the EHL data will be electronically sent to the child's WIC nutritionist, to be read prior to a WIC nutrition appointment with that client.

Information from the WIC nutritionist appointments, including nutrition counseling codes from each appointment in addition to collected health information will then be sent to the child's pediatrician, to be included as part of the child's electronic health record.

Child's growth measures will be taken from the well baby visits, along with any unique information from the WIC nutritionist visits. In addition, data collection surveys will be distributed to all study participants at 2, 5 and 7 months after birth, either electronically or by paper packet.

ELIGIBILITY:
Inclusion Criteria:

* mother is English speaking, infant is a singleton birth, infant birthweight greater than or equal to 2500g, infant gestational age at least 37 weeks, infant no more than 2 months old, no plans for baby to be put up for adoption, no congenital or neonatal conditions that would affect growth, mother has no major morbidities that would affect postpartum care, eligible and/or enrolled in a WIC program in central PA, infant pediatrician is a Geisinger physician in a pediatric service line in Luzerne county

Exclusion Criteria:

* non-English speaking, mother is planning to leave the county where she enrolled within 6-9 months, mother is less than 18 years of age, mother is older than 55 years of age

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 289 (Actual)
Dates: Start 2016-07-06 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Infant Growth Measures | At birth, and approximately at 2, 5 and 7 months after birth
  Weight, length and age of child at each well-child visit, to calculate sex-specific weight-for-age z-scores and percent overweight based on World Health Organization (WHO) standards
Infant rapid weight gain | From birth to 6 months
  Change in sex-specific weight-for-age z-scores from birth to 6 months as described by LJ Griffiths

SECONDARY OUTCOMES:
Changes in attitudes, beliefs, knowledge, and parenting self-efficacy | At approximately 2, 5 and 7 months postpartum
  Through behavioral surveys, the investigators will assess changes in attitudes, knowledge, and beliefs about parenting, and additionally parenting self-efficacy, and consistency of messages will also be assessed
Maternal knowledge/awareness of coordinated care | 7 months postpartum
  Assessed through Perceived Involvement in Care survey
Care coordination between WIC and Geisinger settings | At approximately 2, 5 and 7 months postpartum
  Care coordination between settings will be evaluated by monitoring the secure flow of participant-level data between Geisinger and WIC for data sharing, care coordination opportunities and documented care.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S Savage, PhD, Principal Investigator — Penn State University; Lisa Bailey-Davis, DEd, Study Director — Geisinger Health Systems
Locations (1):
- Geisinger Health Systems, Danville, Pennsylvania, United States

REFERENCES:
- [Derived] Savage JS, Moore AM, Kling SMR, Marini M, Hernandez E, Franceschelli Hosterman J, Hassink S, Paul IM, Bailey-Davis L. Coordination Between Primary Care and Women, Infants, and Children to Prevent Obesity for Infants from Low-Income Families: A Pragmatic Randomized Clinical Trial. Child Obes. 2023 Dec;19(8):515-524. doi: 10.1089/chi.2022.0137. Epub 2022 Nov 11. PMID 36367983
- [Derived] Kling SM, Harris HA, Marini M, Cook A, Hess LB, Lutcher S, Mowery J, Bell S, Hassink S, Hayward SB, Johnson G, Franceschelli Hosterman J, Paul IM, Seiler C, Sword S, Savage JS, Bailey-Davis L. Advanced Health Information Technologies to Engage Parents, Clinicians, and Community Nutritionists in Coordinating Responsive Parenting Care: Descriptive Case Series of the Women, Infants, and Children Enhancements to Early Healthy Lifestyles for Baby (WEE Baby) Care Randomized Controlled Trial. JMIR Pediatr Parent. 2020 Nov 24;3(2):e22121. doi: 10.2196/22121. PMID 33231559
- [Derived] Savage JS, Kling SMR, Cook A, Hess L, Lutcher S, Marini M, Mowery J, Hayward S, Hassink S, Hosterman JF, Paul IM, Seiler C, Bailey-Davis L. A patient-centered, coordinated care approach delivered by community and pediatric primary care providers to promote responsive parenting: pragmatic randomized clinical trial rationale and protocol. BMC Pediatr. 2018 Sep 4;18(1):293. doi: 10.1186/s12887-018-1263-z. PMID 30180831

DOCUMENTS (1):
  • Study Protocol (2018-02-19): https://cdn.clinicaltrials.gov/large-docs/08/NCT03482908/Prot_000.pdf